CLINICAL TRIAL: NCT02701309
Title: Non-invasive Optical Detection of Iron Deficiency in Children- Evaluation of a Fiber Optic Tissue Fluorescence Measurement to Determine the Erythrocyte Zinc Protoporphyrin-IX/Heme Ratio
Brief Title: Non-invasive Optical Detection of Iron Deficiency in Children
Acronym: IronKids
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Koletzko - Office, Prof. Dr., Ludwig-Maximilians - University of Munich
Other Study IDs: LFL_02/2015
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Iron Deficiency; Iron-deficiency Anemia; Child
Keywords: Iron deficiency; Child; Infancy; Preschool children; iron deficiency anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-invasive Iron detection: Children between 9months and 5years will be recruited for a non-invasive iron measurement on the lower lip. This study is focusing on the feasability of a non-invasive detection method. There is no intervention planed. The device is tested once for 3-5 Minutes.
  Interventions: Device: Non-invasive Iron detection device via Zinc-Protoporphyrin

INTERVENTIONS:
Device: Non-invasive Iron detection device via Zinc-Protoporphyrin — In this study the feasability, sensitivity and specifity of a non-invasive detection method of zinc-protoporphyrin in children is evaluated. It´s a one-arm study, without control Group. Children are aged between 9m and 5y and have a clinical blood sampling indicated.
  Other Names: Iron detection device

SUMMARY:
This study aims to evaluate a prototype device detecting zinc protoporphyrin-IX fluorescence non-invasively from the intact oral mucosa in children. The prototype device has shown high sensitivity and specificity in women after delivery for iron deficiency. Children are at increased risk for iron deficiency and prevention methods are not established jet. Zinc protoporphyrin-IX is an early indicator of iron deficiency and may be more sensitive than other established parameters. The prototype device is used to measure the erythrocyte zinc protoporphyrin-IX/heme ratio in children aged 9 months to 5 years. Children in this age are at increased risk for iron deficiency as they are growing rapidly and iron deficiency in this age may affect the neurodevelopment and immune system adversely. It is proposed that these effects cannot be rectified by iron supplementation in later years. The results from the non-invasive measurements are compared to reference measurements of the erythrocyte zinc protoporphyrin-IX/heme ratio from residual blood samples from the same patients and to other indicators of iron status, including hemoglobin, ferritin, serum iron, transferrin, transferrin saturation and soluble transferrin receptor.

DETAILED DESCRIPTION:
This trial is a proof-of-concept study using a prototype fiber optic fluorometer to acquire autofluorescence spectra in children aged 9 months to 5 years and determine the erythrocyte zinc protoporphyrin-IX fluorescence intensity from these spectra. The non-invasively determined fluorescence spectra are evaluated to provide a quantitative measure of the erythrocyte zinc protoporphyrin-IX/heme concentration ratio. These values are primarily compared to an erythrocyte zinc protoporphyrin-IX determined by HPLC from residual blood samples from the same subjects and secondarily to erythrocyte zinc protoporphyrin-IX/heme ratios determined using a commercial hematofluorometer (AVIV, model 206d) and other indicators of iron status, including hemoglobin, ferritin, serum iron, transferrin, transferrin saturation and soluble transferrin receptor

This study could help to establish the non-invasive fluorescence measurement of zinc protoporphyrin-IX as a rapid, easy to use means for point-of-care screening for iron deficiency in resource-limited settings lacking laboratory infrastructure.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9 months to 5 years
* Planed blood sampling, independently from this study
* Informed written consent to participation´s guardian in the study

Exclusion Criteria:

* the ability of the guardian is not given to approve the consent
* transfusion of blood products before entering the study
* blood sampling is not planed for clinical investigations

Ages: 9 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 9 months to 5 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Comparison of non-invasive erythrocyte zinc protoporphyrin IX measurements with HPLC reference (Spearman's Rho correlation, sensitivity and specificity) | 1 day after measurement
  Erythrocyte zinc protoporphyrin IX in the units of μmol/mol heme, as determined from non-invasive fluorescence and remission spectroscopic measurements at the oral mucosa, compared with reference standard determinations of erythrocyte zinc protoporphyrin IX in blood samples by high performance liquid chromatography (HPLC).

SECONDARY OUTCOMES:
Comparison of non-invasive erythrocyte zinc protoporphyrin IX measurements with estimate of body iron (sensitivity and specificity) | 1 day after measurement
  Erythrocyte zinc protoporphyrin IX in the units of μmol/mol heme, as determined from non-invasive fluorescence and remission spectroscopic measurements at the oral mucosa, compared with an estimate of total body iron, determined from the logarithm of the soluble transferrin receptor/ferritin ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof.Dr.med., Principal Investigator — LMU Munich, Germany
Locations (2):
- Germany (2):
  - Div. Metabolic and Nutritional Medicine Dr. von Hauner Children's Hospital Univ. of Munich Medical Centre, Munich, Bavaria
  - LMU Munich, Munich, Bavaria

IPD SHARING:
Plan to Share IPD: Undecided
The principal investigator (PI, Prof. Dr. Dr. B. Koletzko) has access to the study data. The data may be shared with other researchers for specific research purposes if a written request with detailed description of objectives and goals, workplan and statistical analysis plan, strategy to protect data from other uses, publication strategy, and description of the research team and its qualification is provided. Based on the evaluation of proposals, the PI and study team will decided on a case by case basis which data can be provided.